CLINICAL TRIAL: NCT02520531
Title: Scorpio PS vs Scorpio NRG PS - Total Knee Arthroplasty Comparative Investigation of Function
Brief Title: Scorpio Posterior Stabilised (PS) vs Scorpio NRG ("Energize") PS - Total Knee Arthroplasty
Acronym: ScorpioNRGPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20100506 /K-S-006
Record Dates: First submitted 2015-06-11; First posted 2015-08-13 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scorpio PS (Active Comparator): Patients on the waiting list for a total knee prosthesis who fulfil the inclusion and exclusion criteria will be asked to participate in this study and are randomized to receive the Scorpio PS Total Knee Replacement.
  Interventions: Device: Scorpio PS (posterior stable)
- Scorpio NRG PS (Active Comparator): Patients on the waiting list for a total knee prosthesis who fulfil the inclusion and exclusion criteria will be asked to participate in this study and are randomized to receive the Scorpio NRG PS Total Knee Replacement.
  Interventions: Device: Scorpio NRG PS

INTERVENTIONS:
Device: Scorpio PS (posterior stable) — Implantation of total knee prosthesis
  Arms: Scorpio PS
Device: Scorpio NRG PS — Implantation of total knee prosthesis
  Arms: Scorpio NRG PS

SUMMARY:
Single-centre, prospective, randomized comparative study to compare the maximum flexion and Chair Raise achievement ratios of the Scorpio PS and and the Scorpio NRG PS. Documentation of all complications.

DETAILED DESCRIPTION:
Surveillance design: Single-centre, prospective, randomized comparative study. Objectives: To compare the maximum flexion (active and passive) and Chair Raise achievement ratios. All complications will be documented.

Number of subjects to be enrolled: All consecutive Scorpio patients are included until a group size of 88 is reached.

Clinical evaluations: Chair raise test, Stair climb test, Western Ontario McMaster Osteoarthritis Index (WOMAC) patient self evaluation, EuroQuol - 5 dimension (EQ-5D) patient questionnaire. Standard clinical, functional and pain parameters (Knee Society Score), pre-operatively and post-operatively. All per- and post-op complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a primary total knee arthroplasty (TKA)
* Male and nonpregnant female patients
* Between 18 and 80 years of age at time of surgery
* Patients with a diagnosis of osteoarthritis (OA), avascular necrosis (AVN), and not severe posttraumatic arthritis
* No previous osteosynthesis of the involved knee during the last 12 months
* Patients who understand the conditions of the study and are wiling to participate for the length of the described follow up
* Patients who are capable of, and have given, informed consent for participation in the study

Exclusion Criteria:

* Patients requiring revision surgery of a previous implanted total knee system
* Patients with a diagnosis of severe posttraumatic arthritis (TA) and rheumatoid arthritis (RA)
* Patients with active infection
* Patients with malignancy
* Patients with an immobile hip or ankle arthrodesis
* Severe obese patients (BMI > 35)
* Patients with a neurological deficit
* Previous history of unicompartmental knee arthroplasty or patellar prosthesis
* Patients with concurrent illnesses which are likely to affect their outcome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feczko, MD, Principal Investigator — Clinical Trial Center Maastricht BV
Locations (1):
- Central Trial Center Maastricht BV, Maastricht, Limburg, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scorpio PS | Scorpio NRG PS
Started | 42 | 42
Completed | 36 | 36
Not Completed | 6 | 6
Not completed — Revision of study device components | 2 | 2
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Meet exclusion criterion | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not study device | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scorpio PS | Scorpio NRG PS | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 23 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.44 (8.01) | 66.22 (8.09) | 65.83 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 24 | 23 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Maximum Passive and Active Flexion.
Description: Comparison of maximum flexion, both passive and active between Scorpio NRG PS knee prosthesis and the Scorpio PS knee prosthesis.
  The active flexion-tolerated range is greater/equal 70 degree. The passive flexion-tolerated range is greater/equal 80 degree. The Hyperextension tolerated range is 0 to 10 degree. Higher scores mean a better outcome.
Time Frame: 5 years follow-up
Population: At the 5 years follow-up data of 36 participants per study arm were analyzed.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Scorpio PS | Scorpio NRG PS
Number analyzed (Participants) | 36 | 36
degree
  Passive range of motion | 124.58 (10.04) | 125.14 (23.01)
  Passive Flexion | 126.64 (9.22) | 131.33 (8.49)
  Passive Extension | 1.81 (2.33) | 2.72 (2.48)
  Active range of motion | 118.64 (10.15) | 125.72 (8.66)
  Active Extension | 0.61 (1.08) | 0.97 (1.50)
  Active Flexion | 120.11 (9.77) | 126.69 (8.75)

2. Secondary Outcome: Knee Society Score (KSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: pre-operative, 6, 12, 26 weeks and 1, 2 and 5 years follow-up
Population: Because some patients missed to attend some visits as well as early termination cases, the numbers in some follow-ups differ from number analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio PS | Scorpio NRG PS
Number analyzed (Participants) | 42 | 42
units on a scale
  Pain motion Score pre-op | 47.65 (11.18) | 49.85 (15.31)
  Pain motion Score 6 weeks: number analyzed (Participants) | 39 | 42
  Pain motion Score 6 weeks | 61.65 (16.45) | 69.63 (17.22)
  Pain motion Score 12 weeks: number analyzed (Participants) | 38 | 41
  Pain motion Score 12 weeks | 67.66 (13.00) | 75.38 (13.34)
  Pain motion Score 26 weeks: number analyzed (Participants) | 41 | 40
  Pain motion Score 26 weeks | 71.58 (14.61) | 74.70 (14.01)
  Pain motion Score 1 year: number analyzed (Participants) | 39 | 41
  Pain motion Score 1 year | 70.27 (12.39) | 73.83 (13.98)
  Pain motion Score 2 years: number analyzed (Participants) | 37 | 41
  Pain motion Score 2 years | 71.29 (13.96) | 74.79 (12.11)
  Pain motion Score 5 years: number analyzed (Participants) | 36 | 36
  Pain motion Score 5 years | 69.42 (11.94) | 74.85 (11.39)
  Function Score pre-op | 61.55 (12.12) | 60.12 (15.36)
  Function Score 6 weeks: number analyzed (Participants) | 39 | 42
  Function Score 6 weeks | 56.63 (15.83) | 60.83 (19.16)
  Function Score 12 weeks: number analyzed (Participants) | 38 | 41
  Function Score 12 weeks | 73.29 (19.09) | 82.80 (14.88)
  Function Score 26 weeks: number analyzed (Participants) | 41 | 40
  Function Score 26 weeks | 87.93 (15.49) | 90.25 (17.76)
  Function Score 1 year: number analyzed (Participants) | 39 | 41
  Function Score 1 year | 88.46 (14.38) | 94.88 (12.67)
  Function Score 2 years: number analyzed (Participants) | 37 | 41
  Function Score 2 years | 86.79 (22.52) | 95.24 (10.00)
  Function Score 5 years: number analyzed (Participants) | 36 | 36
  Function Score 5 years | 87.92 (22.05) | 95.14 (10.45)

3. Secondary Outcome: Chair Raise Test
Description: A measurement to assess functional lower extremity strength. The participant is seated on a chair. Arms are crossed at the wrists and held against the chest. The participant is instructed to arise from an adjustable chair with the knees in a 90 degree angle (measurement with Goniometer) without using arms.
Time Frame: pre-operative, 6, 12, 26 weeks and 1, 2 and 5 years follow-up
Population: In some cases it was missed to do the Chair rise test.
Measure: Count of Participants; unit: Participants
Arm/Group | Scorpio PS | Scorpio NRG PS
Number analyzed (Participants) | 42 | 42
Participants
  Can arise from chair pre-operative: number analyzed (Participants) | 30 | 37
  Can arise from chair pre-operative | 26 | 30
  Can arise from chair at 6 weeks: number analyzed (Participants) | 39 | 41
  Can arise from chair at 6 weeks | 34 | 37
  Can arise from chair at 12 weeks: number analyzed (Participants) | 41 | 41
  Can arise from chair at 12 weeks | 39 | 39
  Can arise from chair at 26 weeks: number analyzed (Participants) | 41 | 41
  Can arise from chair at 26 weeks | 40 | 38
  Can arise from chair at 1 year: number analyzed (Participants) | 40 | 41
  Can arise from chair at 1 year | 37 | 39
  Can arise from chair at 2 years: number analyzed (Participants) | 40 | 41
  Can arise from chair at 2 years | 39 | 36
  Can arise from chair at 5 years: number analyzed (Participants) | 36 | 36
  Can arise from chair at 5 years | 34 | 34

4. Secondary Outcome: WOMAC Patient Questionnaire
Description: The WOMAC collects information specific to osteoarthritis outcomes. The patient response questionnaire uses a visual analog scale for pain, measuring factors of general pain, stiffness, and function. Each question is scored from 0 to 4 for each set of factors, with 0 indicating no pain, stiffness, or limited in function, and 4 indicating extreme pain stiffness, or limited in function. Total WOMAC scores range from 0 to 96 wit lower values representing better outcomes.
Time Frame: pre-operative, 12, 26 weeks and 1, 2 and 5 years follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio PS | Scorpio NRG PS
Number analyzed (Participants) | 42 | 42
units on a scale
  Total score pre-operative | 49.33 (14.37) | 47.63 (15.84)
  Total score 12 weeks: number analyzed (Participants) | 41 | 41
  Total score 12 weeks | 26.56 (15.53) | 18.69 (15.22)
  Total score 26 weeks: number analyzed (Participants) | 41 | 41
  Total score 26 weeks | 19.95 (16.66) | 20.21 (19.24)
  Total score 1 year: number analyzed (Participants) | 39 | 41
  Total score 1 year | 19.74 (16.68) | 12.98 (13.78)
  Total score 2 years: number analyzed (Participants) | 39 | 41
  Total score 2 years | 18.56 (20.93) | 13.60 (17.32)
  Total score 5 years: number analyzed (Participants) | 36 | 36
  Total score 5 years | 14.44 (15.92) | 12.24 (16.52)

5. Secondary Outcome: EQ-5D (Euro-Quol 5-Dimension) Patient Questionnaire
Description: The EQ-5D is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
Time Frame: pre-operative, 12, 26 weeks and 1, 2 and 5 years follow-up
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio PS | Scorpio NRG PS
Number analyzed (Participants) | 42 | 42
units on a scale
  Pre-operative EQ-5D | 0.60 (0.21) | 0.53 (0.25)
  12 weeks EQ-5D: number analyzed (Participants) | 41 | 41
  12 weeks EQ-5D | 0.76 (0.16) | 0.77 (0.19)
  26 weeks EQ-5D: number analyzed (Participants) | 41 | 41
  26 weeks EQ-5D | 0.76 (0.20) | 0.78 (0.22)
  1 year EQ-5D: number analyzed (Participants) | 40 | 41
  1 year EQ-5D | 0.72 (0.32) | 0.82 (0.19)
  2 years EQ-5D: number analyzed (Participants) | 39 | 41
  2 years EQ-5D | 0.76 (0.28) | 0.81 (0.24)
  5 years EQ-5D: number analyzed (Participants) | 36 | 36
  5 years EQ-5D | 0.77 (0.26) | 0.80 (0.23)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time point of the study related surgery until termination from study latest at the 5 years follow-up.
Description: Definitions do not differ.
Arm/Group | Scorpio PS | Scorpio NRG PS
All-Cause Mortality (participants affected / at risk) | 1/42 | 2/42
Serious Adverse Events (participants affected / at risk) | 10/42 | 13/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scorpio PS (N=42) | Scorpio NRG PS (N=42)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypopharinx Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac Complaints (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Collapse (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Leakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthroscopic Nettoyage of Knee (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Removal of fibrous tissue & blood
Tooth Implant Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal Corpus Alienum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Corpus alienum in abdomen removed via laparoscopy
Knee pain insert revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tibial Component Revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peri Articular Ossification of Hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate Resection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aneurism (Vascular disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Placement of patella prosthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Patella resurfacing (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-06-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02520531/Prot_SAP_000.pdf